CLINICAL TRIAL: NCT04990544
Title: A Randomized, Double-blinded, Placebo-controlled Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of the Recombinant SARS-CoV-2 Vaccine (CHO Cell) for the Prevention of COVID-19 in Adults Aged 18 Years and Above
Brief Title: Phase II Clinical Trial of Recombinant SARS-CoV-2 Spike Protein Vaccine (CHO Cell) for the Prevention of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Walvax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202-COV-1002
Record Dates: First submitted 2021-08-02; First posted 2021-08-04 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Adult Group 2a (Experimental): Adult healthy subjects (18 to 59 years of age, inclusive) receive 202-CoV low adjuvant dose at Day 0 and Day 28
  Interventions: Biological: 202-CoV low adjuvant dose
- Adult Group 2b (Experimental): Adult healthy subjects (18 to 59 years of age, inclusive) receive 202-CoV low antigen dose at Day 0 and Day 28
  Interventions: Biological: 202-CoV low antigen dose
- Adult Group 2c (Experimental): Adult healthy subjects (18 to 59 years of age, inclusive) receive 202-CoV standard dose at Day 0 and Day 28.
  Interventions: Biological: 202-CoV standard dose
- Adult Placebo (Placebo Comparator): Adult healthy subjects (18 to 59 years of age, inclusive) receive 2 doses of placebo (saline) at Day 0 and Day 28
  Interventions: Biological: Placebo
- Elderly Group 2d (Experimental): Adult healthy subjects (60 years of age and above) receive 202-CoV low adjuvant dose at Day 0 and Day 28
  Interventions: Biological: 202-CoV low adjuvant dose
- Elderly Group 2e (Experimental): Adult healthy subjects (60 years of age and above) receive 202-CoV low antigen dose at Day 0 and Day 28
  Interventions: Biological: 202-CoV low antigen dose
- Elderly Group 2f (Experimental): Adult healthy subjects (60 years of age and above) receive 202-CoV standard dose at Day 0 and Day 28
  Interventions: Biological: 202-CoV standard dose
- Elderly Placebo (Placebo Comparator): Adult healthy subjects (60 years of age and above) receive 2 doses of placebo (saline) at Day 0 and Day 28
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: 202-CoV low adjuvant dose — standard dose of 202-CoV with low dose CpG / alum adjuvant
  Arms: Adult Group 2a; Elderly Group 2d
Biological: 202-CoV low antigen dose — low dose of 202-CoV with CpG / alum adjuvant
  Arms: Adult Group 2b; Elderly Group 2e
Biological: 202-CoV standard dose — standard dose 202-CoV with CpG / alum adjuvant
  Arms: Adult Group 2c; Elderly Group 2f
Biological: Placebo — Normal saline solution
  Arms: Adult Placebo; Elderly Placebo

SUMMARY:
The purpose of this double-blind, randomized, controlled study is to assess immunogenicity and safety of 202-CoV at multiple dose levels, administered as 2 injections (i.m) at 28 days apart in adult subjects 18 years of age and above.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-59 years as well as 60 years and above who can provide legal identification (males and females are both required).
* Willing to participate in the study with informed consent prior to screening
* Negative in SARS-CoV-2 IgG and IgM test at screening.
* Women of childbearing potential must be using effective method of birth control for 14 days prior to the enrollment of the study and must agree to continue such precautions during the study until 30 days after the second dose of the study vaccine/placebo.
* Male subjects must agree to employ acceptable contraception from the day of first dose of the study vaccine/placebo until 30 days after the second dose of the study vaccine/placebo.

Exclusion Criteria:

* Confirmed or asymptomatic COVID-19 cases or SARS-CoV-2 infection(had positive in SARS-CoV-2 nucleic acid test or serological test).
* Had a history of traveling or residence in domestic area of high pandemic risk, overseas or epidemic areas, or had a history of contact with confirmed, asymptomatic or suspected COVID-19 cases within the past 14 days;
* History of SARS;
* Received SARS-CoV-2 vaccines for emergency use or approved SARS-CoV-2 vaccines;
* Individuals involving a clinical study within 6 months prior to the screening visit; or planning to participate in another clinical study during study period.
* Individual's systolic blood pressure ≥ 150mmHg and/or diastolic blood pressure ≥ 100mmHg at screening visit
* Axillary temperature >=37.3℃ prior to vaccination
* Individuals in other acute diseases, or in the acute phase of chronic diseases within 3 days prior to the signing of the informed consent form.
* Received immunoglobulin and/or blood product 3 months prior to the first vaccination.
* Presence of uncontrolled chronic pulmonary, cardiovascular, renal, hepatic, neurologic, hematologic or metabolic (including diabetes mellitus) disorders, which would include the potential subject in a high-risk category for SARS-CoV-2 infection and/or its complications as judged by the investigator.
* Individuals with a history of severe allergic reaction (throat swelling, difficult in breath, dyspnea, or shock).
* Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction [e.g., anaphylaxis to any component of the study vaccines (S protein, Aluminum hydroxide, CpG adjuvant).
* Any autoimmune or immunodeficiency disease/condition [e.g. human immunodeficiency virus (HIV) infection, Systemic lupus erythematosus (SLE)]
* Received immunoglobulin, blood-derived products within 3 months prior to the first study vaccination.
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disease, platelet abnormality) obvious bruises or coagulopathy.
* Pregnant women or breastfeeding women.
* According to the judgment of the investigator, subject has or had any other symptoms, medical history and other factors that are not suitable for participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of SARS-CoV-2 neutralising antibodies | 56 days
  Neutralizing antibody activity as detected by neutralization assay expressed as GMTs at multiple time points through Day 56
Seroconversion rate (SCR) of SARS-CoV-2 neutralising antibodies | 56 days
  Neutralizing antibody activity as detected by neutralization assay expressed as seroconversion rate at multiple time points through Day 56
Geometric mean titer (GMT) of serum IgG antibodies | 56 days
  Serum IgG antibody levels specific for the SARS-CoV-2 S protein antigen as detected by ELISA expressed as GMTs at multiple time points through Day 56
Seroconversion rate (SCR) of serum IgG antibodies | 56 days
  Serum IgG antibody levels specific for the SARS-CoV-2 S protein antigen as detected by ELISA expressed as seroconversion rate at multiple time points through Day 56
Geometric mean fold rise (GMFR) of SARS-CoV-2 neutralising antibodies | 56 days
  GMFR in SARS-CoV-2 serum neutralizing titers from before vaccination to each subsequent time point
Geometric mean fold rise (GMFR) of serum IgG antibodies | 56 days
  GMFR of serum IgG antibodies from before vaccination to each subsequent time point

SECONDARY OUTCOMES:
Percentage of participants reporting adverse events (AEs) | From dose 1 through 28 days after the last dose
  Percentage of participants with solicited AEs (local, systemic) for 28 days following each primary vaccination (Days 0, 28) by intensity, relevance.
Percentage of participants reporting solicited AEs | For 7 days after dose 1 and dose 2
  Percentage of participants with solicited AEs (local, systemic) for 7 days following each primary vaccination (Days 0, 28) by intensity, relevance.
Percentage of participants reporting unsolicited AEs | From dose 1 through 28 days after the last dose
  Percentage of participants with unsolicited AEs for 28 days following each vaccination
Percentage of participants reporting serious adverse events (SAEs) | From dose 1 through 12 months after the last dose
  Percentage of participants with SAEs from dose 1 through 12month after last dose vaccination
Percentage of participants reporting adverse events of special interest (AESIs) | From dose 1 through 12 months after the last dose
  Percentage of participants with AESI from dose 1 through 12month after last dose vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangcheng Center for Disease Control and Prevention, Xuchang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu H, Zhou C, An J, Song Y, Yu P, Li J, Gu C, Hu D, Jiang Y, Zhang L, Huang C, Zhang C, Yang Y, Zhu Q, Wang D, Liu Y, Miao C, Cao X, Ding L, Zhu Y, Zhu H, Bao L, Zhou L, Yan H, Fan J, Xu J, Hu Z, Xie Y, Liu J, Liu G. Development of recombinant COVID-19 vaccine based on CHO-produced, prefusion spike trimer and alum/CpG adjuvants. Vaccine. 2021 Nov 26;39(48):7001-7011. doi: 10.1016/j.vaccine.2021.10.066. Epub 2021 Oct 30. PMID 34750014